CLINICAL TRIAL: NCT00375830
Title: Combined 18F-NaF/18F-FDG PET/MRI for Detection of Skeletal Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-03778; 96754 (Other: Stanford University Alternate IRB Approval Number); BONE0001 (Other: OnCore)
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Technetium Tc 99m Medronate; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18; Gadolinium DTPA; gadofosveset trisodium; gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans (Experimental): Preliminary pilot assessment to confirm feasibility & improved diagnostic accuracy of the combined 18F-NaF CT & 18F-FDG PET scan procedures, as compared to the regular medical care procedure, 99mTc MDP bone scans.
  Interventions: Procedure: Bone scan; Drug: 99mTc-methyl diphosphonate; Procedure: Positron Emission Tomography (PET) scan; Drug: 18F-Fludeoxyglucose (18F-FDG); Procedure: Computed Tomography (CT) scan; Drug: 18F-Sodium Fluoride (18F-NaF); Drug: Gadopentetate dimeglumine
- Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans (Experimental): Assessment to define the accuracy of the combined 18F-NaF CT & 18F-FDG PET/CT scan procedures compared to 99mTc MDP bone scan.
  Interventions: Procedure: Bone scan; Drug: 99mTc-methyl diphosphonate; Procedure: Positron Emission Tomography (PET) scan; Drug: 18F-Fludeoxyglucose (18F-FDG); Procedure: Computed Tomography (CT) scan; Drug: 18F-Sodium Fluoride (18F-NaF); Procedure: Whole Body Magnetic Resonance Imaging (WB-MRI) scan; Drug: Gadofosveset; Drug: Gadobutrol
- Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI scan (Experimental): Assessment to define the utility of 18F-NaF & 18F-FDG as the radiolabels in a single combined PET / WB-MRI procedure.
  Interventions: Procedure: Bone scan; Drug: 99mTc-methyl diphosphonate; Procedure: Positron Emission Tomography (PET) scan; Drug: 18F-Fludeoxyglucose (18F-FDG); Drug: 18F-Sodium Fluoride (18F-NaF); Procedure: Whole Body Magnetic Resonance Imaging (WB-MRI) scan; Drug: Gadofosveset; Drug: Gadobutrol

INTERVENTIONS:
Procedure: Bone scan — Scan to diagnose a number of bone conditions including cancer or metastasis
  Other Names: Bone scintigraphy
Drug: 99mTc-methyl diphosphonate — Radiolabel for bone scan procedures
  Other Names: 99mTc-methylene diphosphonate; Technetium 99mTc medronate; 99mTc-MDP; t99-MDP
Procedure: Positron Emission Tomography (PET) scan — Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
Drug: 18F-Fludeoxyglucose (18F-FDG) — Radiolabel for positron emission tomography scan procedures
  Other Names: 2-Deoxy-2-(18F)Fluoro-D-Glucose; 2-F18-Fluoro-2-deoxy-D-glucose; 2-F18-Fluoro-2-deoxyglucose; 18F 2-Fluoro-2-deoxy-D-Glucose; Fludeoxyglucose F-18; Fluorodeoxyglucose F18
Procedure: Computed Tomography (CT) scan — Scan to detect & analyze X-rays
  Other Names: Computerized Axial Tomograph (CAT) scan; Computer-aided Tomography (CAT) scan
  Arms: Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans; Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans
Drug: 18F-Sodium Fluoride (18F-NaF) — Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
  Other Names: 18F-Sodium Fluorine
Procedure: Whole Body Magnetic Resonance Imaging (WB-MRI) scan — Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Scan that uses strong magnetic fields & radio waves to generate images of the organs in the body.
  Arms: Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans; Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI scan
Drug: Gadopentetate dimeglumine — A gadolinium-based contrast agent for MRI
  Other Names: Magnevist
  Arms: Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans
Drug: Gadofosveset — A gadolinium-based contrast agent for MRI
  Other Names: Ablavar
  Arms: Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans; Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI scan
Drug: Gadobutrol — A gadolinium-based contrast agent for MRI
  Other Names: Gadavist
  Arms: Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET scans; Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI scan

SUMMARY:
This clinical trial studies the use of sodium fluorine-18 (18F-NaF) plus fluorine-18 (18F) fluorodeoxyglucose (FDG) positron emission tomography (PET)/ whole body magnetic resonance imaging (WBMRI) to detect skeletal metastases in patients with stage III-IV breast cancer or stage II-IV prostate cancer.

DETAILED DESCRIPTION:
Eligible participants had previously received a bone scan using the radiolabel 99mTc-methyl diphosphonate (t99-MDP) as part of their regular medical care.

18F-NaF and 18F-FDG are radioactive substances (radiolabels) that are absorbed by cancerous cells and allow for the cancer to be found using diagnostic procedures such as positron emission tomography (PET)/ whole body magnetic resonance imaging (WBMRI). PET/WBMRI is a combination procedure that combines the detailed PET images of areas inside the body from PET with the WBMRI scans, and may help find and diagnose skeletal metastases in patients with breast or prostate cancer. It is not yet known whether 18F-NaF/18F-FDG PET/WBMRI is better than standard imaging methods in detecting skeletal metastases.

Eligible participants diagnosed with breast/prostate cancers and who have had 99mTc MDP bone scanning as part of their routine care are recruited and enrolled. Participants then receive an 18F-NaF/18F-FDG positron emission tomography (PET)/ WBMRI combination scan.

The PET/MRI scans will be interpreted by 2 American Board Nuclear Medicine (ABNM)-certified physicians and 2 American Board of Radiology (ABR)-certified radiologists, all with significant clinical experience, who are blinded to the subjects' medical history and the results of other imaging modalities.

The scans will be analyzed and compared against each other, with a consensus read will be obtained for each scan. Characterization of lesions as true-positive, true-negative, false-positive or false-negative will be done through a combination of clinical follow-up, imaging follow-up and/or histopathology findings. An overall diagnosis based on each scan will be determined on a 5-point scale (1=benign, 2=likely benign, 3=uncertain, 4=likely malignant, 5=malignant) to conduct a receiver operating characteristic (ROC) analysis.

If the diagnosis is positive for metastases on any of the scans, the investigator will identify the number of lesions and locations of positivity, and record this information.

Clinical is obtained at about 12 months after the initial scans.

ELIGIBILITY:
All patients were enrolled after receiving a regular medical care bone scan using the radiolabel 99mTc-methyl diphosphonate (t99-MDP).

INCLUSION CRITERIA

* ≥ 18 years old at the time of the drug administration
* ≥ Stage 3 breast cancer OR ≥ stage 2 prostate cancer OR prostate-specific antigen (PSA) > 10 micrograms/L OR recurrent breast or prostate cancer
* Capable of complying with study procedures
* Able to remain still for duration of imaging procedure (about one hour)
* Written informed consent

EXCLUSION CRITERIA

* Pregnant or nursing
* Metallic implants that contraindicate MRI
* Renal function impairment that contraindicates MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iagaru A, Young P, Mittra E, Dick DW, Herfkens R, Gambhir SS. Pilot prospective evaluation of 99mTc-MDP scintigraphy, 18F NaF PET/CT, 18F FDG PET/CT and whole-body MRI for detection of skeletal metastases. Clin Nucl Med. 2013 Jul;38(7):e290-6. doi: 10.1097/RLU.0b013e3182815f64. PMID 23455520
- [Result] Minamimoto R, Loening A, Jamali M, Barkhodari A, Mosci C, Jackson T, Obara P, Taviani V, Gambhir SS, Vasanawala S, Iagaru A. Prospective Comparison of 99mTc-MDP Scintigraphy, Combined 18F-NaF and 18F-FDG PET/CT, and Whole-Body MRI in Patients with Breast and Prostate Cancer. J Nucl Med. 2015 Dec;56(12):1862-8. doi: 10.2967/jnumed.115.162610. Epub 2015 Sep 24. PMID 26405167
- [Result] Iagaru A, Minamimoto R, Jamali M, Barkodhodari A, Gambhir SS, Vasanawala S. Imaging patients with breast and prostate cancers using combined 18F NaF/18F FDG and TOF simultaneous PET/ MRI. EJNMMI Phys. 2015 Dec;2(Suppl 1):A65. doi: 10.1186/2197-7364-2-S1-A65. No abstract available. PMID 26956325
- [Result] Sonni I, Minamimoto R, Baratto L, Gambhir SS, Loening AM, Vasanawala SS, Iagaru A. Simultaneous PET/MRI in the Evaluation of Breast and Prostate Cancer Using Combined Na[18F] F and [18F]FDG: a Focus on Skeletal Lesions. Mol Imaging Biol. 2020 Apr;22(2):397-406. doi: 10.1007/s11307-019-01392-9. PMID 31236756

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans | Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans | Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI Scan
Started | 10 | 30 | 74
Completed | 10 | 30 | 74
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans | Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans | Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI Scan | Total
Number analyzed (Participants) | 10 | 30 | 74 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 16 | 42 | 63
  >=65 years | 5 | 14 | 32 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.8) | 61.6 (13.0) | 62.9 (11.2) | 62.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 15 | 23 | 43
  Male | 5 | 15 | 51 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 6 | 7
  Not Hispanic or Latino | 7 | 28 | 66 | 101
  Unknown or Not Reported | 3 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 5 | 14 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 2 | 2
  White | 5 | 18 | 52 | 75
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 30 | 74 | 114

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 - NaF PET/CT vs 99mTc-MDP Bone Scintigraphy
Description: The medical value of 18F-sodium fluoride (NaF) positron emission tomography / computed tomography (PET/CT) vs 99mTc-methylene diphosphonate (MDP) bone scintigraphy was assessed on the basis of the radiation oncologist's medical assessment of image quality and detected extent of disease, for each participant. Per protocol, the data were collected and the outcome is reported for Cohort 1 only. The outcome is reported as the number of participants for whom the medical value of the image was superior for 18F-NaF vs 99mTc-MDP bone scintigraphy ("18F-NaF > 99mTc-MDP"), the same between both scans ("18F-NaF = 99mTc-MDP"), or inferior for 18F-NaF vs 99mTc-MDP bone scintigraphy ("18F-NaF < 99mTc-MDP").
Time Frame: 30 days
Population: This assessment was conducted only for Cohort 1 as part of the "pilot phase" of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans
Number analyzed (Participants) | 10
Participants
  18F-NaF > 99mTc-MDP | 10
  18F-NaF = 99mTc-MDP | 0
  18F-NaF < 99mTc-MDP | 0

2. Secondary Outcome: Cohort 1 - 18F-NaF PET/CT vs 18F-FDG PET/CT
Description: The medical value of 18F-sodium fluoride (NaF) positron emission tomography / computed tomography (PET/CT) vs 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) was assessed on the basis of the radiation oncologist's medical assessment of image quality and detected extent of disease, for each participant diagnosed with osseous (skeletal) metastases. Per protocol, the data were collected and the outcome is reported for Cohort 1 only. The outcome is reported as the number of participants for whom the medical value of the image was superior for 18-NaF PET/CT compared to 18F-FDG PET/CT, the same between both scans, or inferior for 18-NaF PET/CT compared to 18F-FDG PET/CT. The outcome result is represented as a number without dispersion.
Time Frame: 30 days
Population: This assessment was conducted only for Cohort 1, and only for participants with skeletal metastases, as part of the "pilot phase" of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans
Number analyzed (Participants) | 3
Participants
  18F-NaF > 18F-FDG | 3
  18F-NaF = 18F-FDG | 0
  18F-NaF < 18F-FDG | 0

3. Secondary Outcome: Cohort 1 - Whole-body MRI vs 18F-NaF PET/CT
Description: The medical value of whole body magnetic imaging resonance (WB-MRI) vs 18F-sodium fluoride (NaF) positron emission tomography / computed tomography (PET/CT) was assessed on the basis of which scan detected the greater number of tumor lesions in each participant. Per protocol, the data were collected and the outcome is reported for Cohort 1 only. The outcome is reported as the number of participants for whom lesions detected by WB MRI was > 18F-NaF PET/CT; equal to 18F-NaF PET/CT; or < 18F-NaF PET/CT. The outcome result is represented as a number without dispersion.
  8 analyzed 5 2
  1
Time Frame: 30 days
Population: This assessment was conducted only for Cohort 1 as part of the "pilot phase" of the study. Only participants with medically-evaluable results for both scans are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans
Number analyzed (Participants) | 8
Participants
  WB MRI > 18F NaF PET/CT | 5
  WB MRI = 18F NaF PET/CT | 2
  WB MRI < 18F NaF PET/CT | 1

4. Secondary Outcome: Cohort 1 - Whole-body MRI vs 18F-FDG PET/CT
Description: The medical value of whole body magnetic imaging resonance (WB-MRI) vs 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) was assessed on the basis of which scan detected the greater number of tumor lesions in each participant. Per protocol, the data were collected and the outcome is reported for Cohort 1 only. The outcome is reported as the number of participants for whom lesions detected by WB MRI was > 18F-FDG PET/CT; equal to to 18F-FDG PET/CT; or < 18F-FDG PET/CT. The outcome result is represented as a number without dispersion.
Time Frame: 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans
Number analyzed (Participants) | 9
Participants
  WB MRI > 18F-FDG PET/CT | 0
  WB MRI = 18F-FDG PET/CT | 6
  WB MRI < 18F-FDG PET/CT | 3

5. Secondary Outcome: Cohort 1 - Detection of Osseous (Skeletal) Metastases by 18F-NaF and 18F-FDG PET/CT
Description: The ability of 18F-sodium fluoride (NaF) and 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) to detect osseous (skeletal) metastases was assessed. Per protocol, the data were collected and the outcome is reported for Cohort 1 only. The outcome is reported as the number of Cohort 1 participants for whom osseous metastases were detected, a number without dispersion.
Time Frame: 30 days
Population: This assessment was conducted only for Cohort 1 as part of the "pilot phase" of the study. Only participants with both medically-evaluable scans are included.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Pilot - 18F-NaF-CT Scan: Preliminary pilot assessment to confirm feasibility & improved diagnostic accuracy of the 18F-NaF CT & 18F-FDG PET scan procedures.
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  Computed Tomography (CT) scan: Scan to detect & analyze X-rays
  18F-Sodium Fluoride (18F-NaF): Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
- Cohort 1 Pilot - 18F-FDG-PET Scan: Preliminary pilot assessment to confirm feasibility & improved diagnostic accuracy of the 18F-NaF CT & 18F-FDG PET scan procedures.
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  18F-Fludeoxyglucose (18F-FDG): Radiolabel for positron emission tomography scan procedures
  Computed Tomography (CT) scan: Scan to detect & analyze X-rays
Arm/Group | Cohort 1 Pilot - 18F-NaF-CT Scan | Cohort 1 Pilot - 18F-FDG-PET Scan
Number analyzed (Participants) | 9 | 9
Participants
  Participants with lesions detected by 18F-NaF | 9 | 6
  Participants with lesions not detected by 18F-NaF | 0 | 3

6. Secondary Outcome: Cohort 2 - 18F-NaF/18F-FDG PET/CT vs Whole-body MRI for Detection of Extraskeletal Lesions
Description: Sensitivity; positive predictive value (PPV); and accuracy for the detection of extraskeletal lesions was assessed for 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) and for whole body magnetic imaging resonance (WB-MRI).
  * Sensitivity is a percentage that defines the proportion of true positive participants with the disease in a total group of participants.
  * PPV is the probability that participants with a positive screening test truly have the disease.
  * Accuracy is the proportion of true results (both true positives and true negatives) among the total number of cases examined.
  Per protocol, the data were collected and the outcome is reported for Cohort 2 only. Sensitivity, PPV, and accuracy are reported as a percentage, a number without dispersion. Higher numbers represent better detection.
Time Frame: 30 days
Population: For this outcome, participants in Cohort 2 were analyzed with 2 distinct scanning procedures, ie, 18F-NaF/18F-FDG PET/CT scan and whole-body MRI scan.
Measure: Number; unit: percentage of particpants
Groups:
- Cohort 2 - Combined 18F-NaF-CT/18F-FDG-PET Scan: Assessment to define the utility of the combined 18F-NaF & 18F-FDG PET/CT scan.
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  18F-Fludeoxyglucose (18F-FDG): Radiolabel for positron emission tomography scan procedures
  18F-Sodium Fluoride (18F-NaF): Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
- Cohort 2 - Whole Body-MRI Scan: Assessment to define the accuracy of the whole body-MRI scan.
  Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Scan that uses strong magnetic fields & radio waves to generate images of the organs in the body.
  Gadofosveset: A gadolinium-based contrast agent for MRI
  Gadobutrol: A gadolinium-based contrast agent for MRI
Arm/Group | Cohort 2 - Combined 18F-NaF-CT/18F-FDG-PET Scan | Cohort 2 - Whole Body-MRI Scan
Number analyzed (Participants) | 30 | 30
percentage of particpants
  Sensitivity | 92.9 | 92.9
  Positive predictive value | 81.3 | 86.7
  Accuracy | 76.5 | 82.4

7. Secondary Outcome: Cohort 2 - 18F-NaF/18F-FDG vs Whole-body MRI for Detection of Skeletal Lesions
Description: Sensitivity and accuracy for the detection of skeletal lesions was assessed for 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) and for whole body magnetic imaging resonance (WB-MRI). Per protocol, the data were collected and the outcome is reported for Cohort 2 only. Sensitivity and accuracy are reported as a percentage, a number without dispersion. Higher numbers represent better detection.
Time Frame: 30 days
Population: as for outcome 6
Measure: Number; unit: percentage of particpants
Groups:
- Cohort 2 - Combined 18F-NaF-CT/18F-FDG-PET Scan: Assessment to define the accuracy of the combined 18F-NaF CT & 18F-FDG PET/CT scan.
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  Computed Tomography (CT) scan: Scan to detect & analyze X-rays
  18F-Fludeoxyglucose (18F-FDG): Radiolabel for positron emission tomography scan procedures
  18F-Sodium Fluoride (18F-NaF): Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
- Cohort 2 - WB-MRI Scan: Assessment to define the accuracy of the whole body MRI scan.
  Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Scan that uses strong magnetic fields & radio waves to generate images of the organs in the body.
  Gadofosveset: A gadolinium-based contrast agent for MRI
  Gadobutrol: A gadolinium-based contrast agent for MRI
Arm/Group | Cohort 2 - Combined 18F-NaF-CT/18F-FDG-PET Scan | Cohort 2 - WB-MRI Scan
Number analyzed (Participants) | 30 | 30
percentage of particpants
  Sensitivity | 96.2 | 81.4
  Accuracy | 89.8 | 74.7

8. Secondary Outcome: Cohort 2 - 18F-NaF/18F-FDG vs 99mTc-MDP Bone Scintigraphy for Detection of Skeletal Lesions
Description: Sensitivity and accuracy for the detection of skeletal lesions was assessed for 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) and for 99mTc-methylene diphosphonate (MDP) bone scintigraphy. Per protocol, the data were collected and the outcome is reported for Cohort 2 only. Sensitivity and accuracy are reported as a percentage, a number without dispersion. Higher numbers represent better detection.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2 Combined 18F-NaF-CT/18F-FDG-PET Scan: Assessment to define the accuracy of the combined 18F-NaF CT & 18F-FDG PET/CT scan procedures.
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  Computed Tomography (CT) scan: Scan to detect & analyze X-rays
  18F-Fludeoxyglucose (18F-FDG): Radiolabel for positron emission tomography scan procedures
  18F-Sodium Fluoride (18F-NaF): Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
- Cohort 2 - 99mTc-MDP Bone Scintigraphy Scan: Assessment to define the utility of the 99mTc-methyl diphosphonate (MDP) bone scintigraphy scan procedure.
  Bone scan: Scan to diagnose a number of bone conditions including cancer or metastasis
  99mTc-methyl diphosphonate: Radiolabel for bone scan procedures
Arm/Group | Cohort 2 Combined 18F-NaF-CT/18F-FDG-PET Scan | Cohort 2 - 99mTc-MDP Bone Scintigraphy Scan
Number analyzed (Participants) | 30 | 30
percentage of participants
  Sensitivity | 96.2 | 64.6
  Accuracy | 89.8 | 65.9

9. Secondary Outcome: Cohort 2 - Overall Sensitivity and Accuracy for 18F-NaF/18F-FDG vs Whole-body MRI
Description: Overall sensitivity and accuracy for the detection of tumor lesions was assessed for 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) and for whole body magnetic imaging resonance (WB-MRI). Per protocol, the data were collected and the outcome is reported for Cohort 2 only. Sensitivity and accuracy are reported as a percentage, a number without dispersion. Higher numbers represent better detection.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2 - Combined 18F-NaF-CT/18F-FDG-PET Scan: Assessment to define the accuracy of the combined 18F-NaF CT & 18F-FDG PET/CT scan procedure;
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  Computed Tomography (CT) scan: Scan to detect & analyze X-rays
  18F-Fludeoxyglucose (18F-FDG): Radiolabel for positron emission tomography scan procedures
  18F-Sodium Fluoride (18F-NaF): Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
- Cohort 2 - Whole Body Magnetic Resonance Imaging (WB-MRI) Scan: Assessment to define the accuracy of the whole body magnetic resonance imaging (WB-MRI) scan procedure.
  Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Scan that uses strong magnetic fields & radio waves to generate images of the organs in the body.
  Gadofosveset: A gadolinium-based contrast agent for MRI
  Gadobutrol: A gadolinium-based contrast agent for MRI
Arm/Group | Cohort 2 - Combined 18F-NaF-CT/18F-FDG-PET Scan | Cohort 2 - Whole Body Magnetic Resonance Imaging (WB-MRI) Scan
Number analyzed (Participants) | 30 | 30
percentage of participants
  Sensitivity | 95.7 | 83.3
  Accuracy | 87.6 | 76.0

10. Secondary Outcome: Cohort 2 - Overall Sensitivity and Accuracy for 18F-NaF/18F-FDG vs Whole-body MRI/99mTc-MDP Bone Scintigraphy
Description: Overall sensitivity and accuracy for the detection of tumor lesions was assessed for 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / computed tomography (PET/CT) and for 99mTc-methylene diphosphonate (MDP) bone scintigraphy. Per protocol, the data were collected and the outcome is reported for Cohort 2 only. Sensitivity and accuracy are reported as a percentage, a number without dispersion. Higher numbers represent better detection.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2 Combined 18F-NaF-CT/18F-FDG-PET Scan: Assessment to define the accuracy of the combined 18F-NaF CT & 18F-FDG PET/CT scan procedure.
  Positron Emission Tomography (PET) scan: Scan to detect gamma rays emitted by a positron-emitting radioligand such as 18F
  Computed Tomography (CT) scan: Scan to detect & analyze X-rays
  18F-Fludeoxyglucose (18F-FDG): Radiolabel for positron emission tomography scan procedures
  18F-Sodium Fluoride (18F-NaF): Radiolabel for CT and PET scans, & as a contrast agent for MRI scans.
- Cohort 2 WB-MRI & 99mTc-MDP Bone Scintigraphy: Assessment to define the accuracy of the 99mTc-methyl diphosphonate (MDP) bone scan procedure.
  Bone scan: Scan to diagnose a number of bone conditions including cancer or metastasis
  99mTc-methyl diphosphonate: Radiolabel for bone scan procedures
Arm/Group | Cohort 2 Combined 18F-NaF-CT/18F-FDG-PET Scan | Cohort 2 WB-MRI & 99mTc-MDP Bone Scintigraphy
Number analyzed (Participants) | 30 | 30
percentage of participants
  Sensitivity | 95.7 | 91.6
  Accuracy | 87.6 | 83.0

11. Secondary Outcome: Cohort 3 - Skeletal Lesions Identified by 99mTc MDP WBBS vs 18F-NaF / 18F-FDG PET/MRI
Description: Participants in Cohort 3 received 99mTc-methylene diphosphonate (MDP) whole-body bone scintigraphy (WBBS) and 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / magnetic imaging resonance (PET/MRI) scans. On the basis of the scans, participants with skeletal lesions were identified. The outcome is reported as the number of Cohort 3 participants for whom skeletal lesions were identified by each scan methodology, a number without dispersion.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3 - 99mTc-methyl Diphosphonate (MDP) Bone Scan: Assessment to define the utility of 99mTc-methyl diphosphonate (MDP) whole-body bone scintigraphy (WBBS)
  Bone scan: Scan to diagnose a number of bone conditions including cancer or metastasis
  99mTc-methyl diphosphonate: Radiolabel for bone scan procedures
- Cohort 3 - 18F-NaF / 18F-FDG PET/MRI: Assessment to define the utility of 18F-NaF & 18F-FDG as the radiolabels in a single combined PET / WB-MRI procedure.
  Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Whole Body Magnetic Resonance Imaging (WB-MRI) scan: Scan that uses strong magnetic fields & radio waves to generate images of the organs in the body.
  Gadofosveset: A gadolinium-based contrast agent for MRI
  Gadobutrol: A gadolinium-based contrast agent for MRI
Arm/Group | Cohort 3 - 99mTc-methyl Diphosphonate (MDP) Bone Scan | Cohort 3 - 18F-NaF / 18F-FDG PET/MRI
Number analyzed (Participants) | 74 | 74
Participants | 37 | 45

12. Secondary Outcome: Cohort 3 - Total Skeletal Lesions Identified, Tc-99m MDP WBBS vs 18F-NaF / 18F-FDG PET/MRI
Description: Participants in Cohort 3 received 99mTc-methylene diphosphonate (MDP) whole-body bone scintigraphy (WBBS) and 18F-sodium fluoride (NaF) / 18F-fluorodeoxyglucose (FDG) positron emission tomography / magnetic imaging resonance (PET/MRI) scans. On the basis of the scans, the total number skeletal lesions identified in the participants was determined. The outcome is reported as the total number skeletal lesions identified by each scan methodology, a number without dispersion.
Time Frame: 30 days
Measure: Number; unit: lesions
Arm/Group | Cohort 3 - 99mTc-methyl Diphosphonate (MDP) Bone Scan | Cohort 3 - 18F-NaF / 18F-FDG PET/MRI
Number analyzed (Participants) | 74 | 74
lesions | 81 | 140

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cohort 1 Pilot-WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans | Cohort 2 WB-MRI & Combined 18F-NaF-CT/18F-FDG-PET Scans | Cohort 3 Combined 18F-NaF / 18F-FDG PET/WB-MRI Scan
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/30 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 0/74
Other Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT00375830/Prot_SAP_001.pdf